CLINICAL TRIAL: NCT05249088
Title: Protocolized Reduction of Non-resuscitation Fluids Versus Usual Care in Septic Shock Patients: A Multicentre Feasibility Trial
Brief Title: Protocolized Reduction of Non-resuscitation Fluids vs Usual Care in Septic Shock Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: REDUSE feasibility trial
Record Dates: First submitted 2022-02-08; First posted 2022-02-21 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-10

CONDITIONS: Shock, Septic
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The clinical team caring for participants will not be blinded due to nature of the intervention. The participants, their family and health personnel responsible for outcome assessment at follow-up will be blinded to the allocation of the intervention. The steering group, author group, trial statistician, outcome assessors, prognosticators, statisticians, and the trial coordinating team will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocolised reduction of non-resuscitation fluids (Experimental): Participants receive non-resuscitation fluids according to a pre-defined protocol starting within two hours of randomization. The intervention is continued for the duration of the ICU admission up to a maximum of 90 days.
  Interventions: Other: Protocolised reduction of non-resuscitation fluids
- Usual Care (Other): Participants receive non-resuscitation fluids according to local routines.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Protocolised reduction of non-resuscitation fluids — * Maintenance fluids are discontinued in participants with positive cumulative fluid balance who are not dehydrated
  * Intravenous fluid and enteral water are given as needed to correct electrolyte disturbances
  * Enteral nutrition with energy density of at least 2 kcal/ml is administered according to local practice
  * Starting 72 hours after inclusion, glucose at a concentration of at least 20% and a maximal dose of 1g/kg/day may be used as nutrition if enteral feeding is not tolerated. Glucose at this dose or lower may be started earlier in patients with insulin dependent diabetes if enteral feeding is not tolerated and local protocol mandates this
  * Parenteral nutrition is administered according to local protocol
  * Intravenous medications are concentrated according to a predefined protocol
  * Patients with neutral or negative cumulative fluid balance receive maintenance and other fluids such that total dose of fluids covers the daily need of water (about 1ml/kg/h)
  Arms: Protocolised reduction of non-resuscitation fluids
Other: Usual care — Participants receive non-resuscitation fluids according to local routines, with the following stipulations:
  * Maintenance fluids (crystalloids and/or glucose and/or enteral water) are given at a dose of 1 ml/kg/h unless local protocol states otherwise
  * Glucose is used at maximal concentration of 10% unless local protocol states otherwise.
  * Medications are concentrated according to local protocol
  Arms: Usual Care

SUMMARY:
The objectives of this feasibility trial are to assess the efficacy and feasibility of methods and procedures of a protocol purposed to compare a reduction of administration of non-resuscitation fluids to usual care in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age)
* Septic shock according to the Sepsis 3 criteria: suspected or confirmed infection AND infusion of vasopressor/inotrope to maintain mean arterial pressure of 65 mmHg or above despite adequate fluid resuscitation AND lactate of 2 mmol/L or above at any time following ICU admission when there was a simultaneous need for vasopressor/inotrope.
* Inclusion within 12 hours after ICU admission.

Exclusion Criteria:

* Confirmed or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Difference in fluid administration | Within the first three days after inclusion (days 0-3)
  Total difference in litres of administered fluids between groups

SECONDARY OUTCOMES:
Proportion of participants with sufficient clinical outcome data | Within 90 days after inclusion
  Fraction of randomised patients with sufficient data for the following clinical outcomes: all-cause mortality, days alive and free of mechanical ventilation, acute kidney injury, and ischemic events in the ICU (cerebral, cardiac, intestinal or limb ischemia)
Proportion of participants assessed by EQ5D-5L and MoCA | 6 months after inclusion
  Fraction of surviving randomized patients who were assessed by European Quality of Life-5 Dimensions 5- Level questionnaire (EQ5D-5L) and The Montreal Cognitive Assessment (MoCA)
Inclusion of eligible patients | During inclusion
  Fraction of all eligible patients who were randomised and consented
Protocol violations | Within 90 days after inclusion
  Fraction of patients experiencing at least one protocol violation

OTHER OUTCOMES:
Mortality | 90 days after inclusion
  All-cause mortality
Complications in the ICU | from randomization until final discharge from ICU or death, whichever comes first, assessed up to 90 days
  Number of patients with one or more of the following complications in the ICU: cerebral, cardiac, intestinal or limb ischemia, or any acute kidney injury
Days alive and free of mechanical ventilation | Within 90 days after inclusion
  Days alive and free of mechanical ventilation
Cognitive function | 6 months after inclusion
  Cognitive function measured using MoCA
Health-Related Quality of Life | 6 months after inclusion
  Health-Related Quality of Life measured using the EQ5D-5L questionnaire
Total volume of non-resuscitation fluids administered | Within the first three days (days 0-3) and within the first five days (days 0-5) after inclusion
  Total volume of non-resuscitation fluids administered
Renal function | Within 90 days after inclusion
  Acute kidney injury stages according to Kidney Disease Improving Global Outcomes [KDIGO] criteria, urea, and days alive and free of renal replacement therapy [RRT]
Gastrointestinal function | Within 90 days after inclusion
  Days alive with full enteral nutrition
Total volume of resuscitation fluids administered | Within the first three days (days 0-3) and within the first five days (days 0-5) after inclusion
  Total volume of resuscitation fluids administered
Cumulative fluid balance | On day 3 and day 5 after inclusion
  Cumulative fluid balance (excluding evaporation)
Diuretics administered | Within the first five days (days 0-5) after inclusion
  Daily dose and type of diuretics administered
Hemodynamic stability | Within the first five days (days 0-5) after inclusion
  Daily highest dose of noradrenaline, daily lactate, and cardiovascular sequential organ failure assessment [SOFA] score
Ischemic events | from randomization until final discharge from ICU or death, whichever comes first, assessed up to 90 days
  Number of patients with one or more ischemic events while in the ICU (cerebral, cardiac, intestinal or limb ischemia)
GOSE score | 6 months after inclusion
  Glasgow Outcome Scale Extended (GOSE) score

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bentzer, MD, PhD, Principal Investigator — Region Skåne
Locations (8):
- Sweden (8):
  - Sahlgrenska University Hospital, Gothenburg
  - Halmstad Hospital, Halmstad
  - Helsingborg Hospital, Helsingborg
  - Kristianstad Hospital, Kristianstad
  - Skåne University Hospital, Lund, Lund
  - Skåne University Hospital, Malmö, Malmo
  - Östersund Hospital, Östersund
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Beginning 9 months after publication of the main report of this trial individual de-identified data will be available for sharing with researchers who provide a methodologically sound proposal as judged by the steering committee. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Linden A, Fisher J, Lilja G, Olsen MH, Sjovall F, Jungner M, Spangfors M, Samuelsson L, Oras J, Linder A, Unden J, Kander T, Lipcsey M, Nielsen N, Jakobsen JC, Bentzer P. Protocolised reduction of non-resuscitation fluids versus usual care in patients with septic shock (REDUSE): a protocol for a multicentre feasibility trial. BMJ Open. 2023 Feb 28;13(2):e065392. doi: 10.1136/bmjopen-2022-065392. PMID 36854601
- [Derived] Linden A, Spangfors M, Olsen MH, Fisher J, Lilja G, Sjovall F, Jungner M, Lengquist M, Kander T, Samuelsson L, Johansson J, Palmnas E, Unden J, Oras J, Cronhjort M, Chew M, Linder A, Lipcsey M, Nielsen N, Jakobsen JC, Bentzer P; REDUSE Trial Group. Protocolized reduction of non-resuscitation fluids versus usual care in septic shock patients (REDUSE): a randomized multicentre feasibility trial. Crit Care. 2024 May 17;28(1):166. doi: 10.1186/s13054-024-04952-w. PMID 38760833
- See also: Markus Harboe Olsen, et al. Protocolised Reduction of Non-resuscitation Fluids Versus Usual Care in Septic Shock Patients (REDUSE) - a Statistical Analysis Plan for a Multicentre Feasibility Trial. 3.00, Zenodo, Dec. 2022, doi:10.5281/zenodo.7392132. — https://zenodo.org/records/7392132